CLINICAL TRIAL: NCT00057291
Title: Effect of Improving Caregiving on Early Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 5R01HD39017-2; 5R01HD039017 (NIH)
Record Dates: First submitted 2003-03-31; First posted 2003-04-01 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2004-12

CONDITIONS: Child Development Disorders
Keywords: Orphanage; Caregiving; Training; Child development
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- caregiving intervention (Experimental): One group received caregiving intervention, another received only training, and a third was business as usual. These were the interventions.
  Interventions: Behavioral: Responsive caregiving

INTERVENTIONS:
Behavioral: Responsive caregiving — Responsive caregiving consisted of operational circumstances and training of caregivers.

SUMMARY:
This study evaluates the effect on children and caregivers of providing training in warm, sensitive, responsive caregiving to caregivers in three orphanages in St. Petersburg, Russia. The study also assesses the effectiveness of having more consistent care from fewer caregivers in a family-like environment.

DETAILED DESCRIPTION:
This project will provide experimental evidence that warm, sensitive, responsive caregiving and structural changes that promote more consistent and fewer caregivers will lead to better physical, mental, social, and emotional development of young children. Structural changes are designed to facilitate a more family-like environment and include smaller group sizes, more consistent caregiving from fewer caregivers, integration by age and disability status, and establishing two daily 60-minute Family Hours in which children and caregivers interact together. The project also attempts to demonstrate that training caregivers can be beneficial to both caregivers and children.

All caregivers and children in three orphanages for children under 4 years old in St. Petersburg, Russia will participate in this study. One orphanage will implement both training and structural changes. A second orphanage will receive training only. The third orphanage will serve as a control, receiving neither training nor structural changes. Caregivers are assessed annually for attitudes to and problems with their jobs; anxiety and depression; coping styles; traditional versus progressive attitudes toward caregiving; sensitivity to children's emotions; values; and perceptions of their own relationships. Children are assessed at 3, 6, 9, 12, 18, 24, 36, and 48 months for physical growth, chronic and acute disorders, functional abilities, and mental, motor, social, and emotional development.

ELIGIBILITY:
Inclusion Criteria

* All caregivers and children in three Baby Homes in St. Petersburg, Russia, who remain in the Baby Homes for at least 4 months.

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1521 (Actual)
Dates: Start 2000-04; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
children's physical growth | 4 to 9+ months
  Improved physical growth
Children's development (mental, motor, social and emotional) | 4 to 9+ months
  Improved behavioral development

CONTACTS AND LOCATIONS:
Overall Officials: Robert B. McCall, Principal Investigator — University of Pittsburgh
Locations (1):
- Baby Home #13, Saint Petersburg, Canal Gnboedora 98, Russia